CLINICAL TRIAL: NCT07186166
Title: Lateral Window Sinus Augmentation in Severe Maxillary Atrophy: A Histological and Histomorphometric Study Using Allograft and Bone Substitute
Brief Title: Sinus Augmentation With Allograft-Bone Substitute in Severe Maxillary Atrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Can Tho University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CTUMP
Record Dates: First submitted 2025-08-30; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Implant Site Reaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lateral Window Sinus Floor Augmentation with 30% HA + 70% β-TCP Graft (Experimental): A prospective single-arm clinical trial was conducted on 60 posterior maxillary edentulous sites in 42 patients with residual bone height < 4 mm. All sites underwent LWSFA, followed by grafting with a 1:1 ratio of 30% HA and 70% β-TCP. At 6 months post-operation, core biopsies were collected during implant placement for histologic evaluation of the grafted sites.
  Interventions: Combination Product: 30% HA+70% β-TCP (Osteon II, Dentium, Korea)

INTERVENTIONS:
Combination Product: 30% HA+70% β-TCP (Osteon II, Dentium, Korea) — A prospective analysis was performed on a single-arm clinical trial involving 60 posterior maxillary edentulous sites in 42 patients with a residual bone height of <4 mm. All sites were treated with lateral window sinus floor augmentation (LWSFA), followed by grafting using a 1:1 ratio of 30% HA with 70% β-TCP (Osteon II, Dentium, Korea). At 6 months postoperatively, core biopsies were harvested during implant placement to assess the histological outcomes of the grafted sites.

SUMMARY:
This study was conducted in two phases. In Phase 1, lateral window sinus floor augmentation was performed using a mixture of hydroxyapatite (30%) and β-tricalcium phosphate (70%) combined with autologous platelet-rich fibrin (PRF). Standard surgical protocols were followed, including prophylactic antibiotics, local anesthesia, and careful elevation of the Schneiderian membrane prior to graft placement.

In Phase 2, after six months of healing, core bone biopsies were harvested with a trephine drill at the planned implant site for histological analysis. Specimens were processed using standardized laboratory protocols and evaluated with light microscopy and digital imaging. Quantitative histomorphometric analysis was performed using ImageJ software to determine the area fractions of newly formed bone and residual graft material. Following biopsy retrieval, dental implants were placed and primary stability was measured with the Implant Stability Quotient (ISQ).

DETAILED DESCRIPTION:
Phase 1: Lateral window sinus floor augmentation, bone graft The patient was prescribed a prophylactic antibiotic regimen consisting of Amoxicillin with Clavulanic Acid (1 g Augmentin tablet), taken one hour before the procedure. Local anesthesia was administered using 2% Lidocaine with Epinephrine (1:100,000). A crestal incision was made along the maxillary alveolar ridge, and a full-thickness mucoperiosteal flap was elevated to expose the surgical site. A lateral window was then prepared in the lateral maxillary wall using a piezotome. The Schneiderian membrane was carefully elevated using the sinus lift augmentation technique. For the grafting procedure, the material was prepared by mixing 30% HA with 70% β-TCP (Osteon II, Dentium, Korea), in a 1:1 ratio, combined with autologous Platelet-Rich Fibrin (PRF) obtained from the patient's blood.

Phase 2: The histological analysis of the bone grafts and implant placement After a healing period of six months, a second-stage surgery was carried out to remove bone tissue and place the implant. At the designated implant site, a trephine drill with a 3 mm outer diameter was used to obtain a core bone biopsy specimen for histological analysis. The biopsy samples were encoded, fixed in 10% formalin, and submitted to the Embryology Department at the University of Medicine and Pharmacy at Ho Chi Minh City, where a standardized protocol was followed for specimen preparation. Histological evaluation was performed using an Olympus BX51 optical microscope connected to an Olympus DP72 12.5 MP digital camera, with captured images transmitted to a computer for assessment of histological parameters. Following biopsy retrieval, the implant osteotomy was completed, and the implant was inserted. Primary stability was assessed using the Implant Stability Quotient (ISQ) index.

Histological sections were analyzed using ImageJ software to quantify the area fractions of newly formed bone and residual graft particles, following established protocols. For each biopsy, three stained sections were evaluated, and the mean value was calculated. The regions corresponding to newly formed bone and residual graft material were delineated using the polygon selection tool, and the software computed their surface areas. The area fraction percentage (AA%) was then expressed as a proportion of the total image surface.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a residual bone height ≤4 mm
* minimum prosthetic space of 5 mm

Exclusion Criteria:

* Patients with acute or chronic maxillary sinusitis, bleeding disorders, diabetes mellitus, bone metabolic diseases, periodontal disease, or malignancies were excluded.
* taking medications that could affect bone metabolism or hemostasis
* Smokers and pregnant women were also excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Histological outcomes | Baseline (T0), After 6 months (T6)
  Histomorphometric evaluation of core biopsies obtained 6 months after maxillary sinus augmentation to quantify the percentage of newly formed bone, residual graft material, and connective tissue. Data will be summarized as mean ± SD and compared between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Can Tho University of Medicine and Pharmacy, Can Tho, Vietnam

IPD SHARING:
Plan to Share IPD: No